CLINICAL TRIAL: NCT02943577
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study of Rapastinel as Adjunctive Therapy in Major Depressive Disorder
Brief Title: A Study of Rapastinel as Adjunctive Therapy in Major Depressive Disorder (RAP-MD-03)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAP-MD-03
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Results first posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — GLYX-13 peptide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rapastinel 450 mg (Experimental): Rapastinel 450 mg weekly intravenous (IV) injections. Each participant will continue to take the same dose of antidepressant therapy the participant was receiving prior to entering this study throughout treatment.
  Interventions: Drug: Rapastinel
- Placebo (Placebo Comparator): Placebo-matching rapastinel weekly IV injections. Each participant will continue to take the same dose of antidepressant therapy the participant was receiving prior to entering this study throughout treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rapastinel — Rapastinel pre-filled syringes for weekly IV injections.
  Arms: Rapastinel 450 mg
Drug: Placebo — Placebo-matching rapastinel pre-filled syringes for weekly IV injections.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy, safety, and tolerability of rapastinel 450 milligrams (mg) compared to placebo adjunctive to antidepressant therapy (ADT) in patients with major depressive disorder (MDD) who have a partial response to ADT.

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for MDD
* Current major depressive episode of at least 8 weeks and not exceeding 18 months in duration at Visit 1
* Have no more than partial response (< 50% improvement) to ongoing treatment with a protocol-allowed antidepressant
* If female of childbearing potential, have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test.

Exclusion Criteria:

* DSM-5-based diagnosis of any disorder other than MDD that was the primary focus of treatment within 6 months before Visit 1
* Lifetime history of meeting DSM-5 criteria for:

  1. Schizophrenia spectrum or other psychotic disorder
  2. Bipolar or related disorder
  3. Major neurocognitive disorder
  4. Neurodevelopmental disorder of greater than mild severity or of a severity that impacts the participant's ability to consent, follow study directions, or otherwise safely participate in the study
  5. Dissociative disorder
  6. Posttraumatic stress disorder
  7. MDD with psychotic features
* Significant suicide risk, as judged by the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Hoogerheyde, Study Director — Allergan
Locations (40):
- United States (40):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - NoesisPharma, Phoenix, Arizona
  - Sun Valley Research Center, Imperial, California
  - Irvine Center for Clinical Research, Inc, Irvine, California
  - NRC Research Institute, Orange, California
  - Asclepes Research Centers, Panorama City, California
  - Artemis Institute for Clinical Research, San Marcos, California
  - MCB Clinical Research Center, Colorado Springs, Colorado
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Research Centers of America, Hollywood, Florida
  - Innova Clinical Trials Inc., Miami, Florida
  - Combined Research Orlando Phase I-IV, Orlando, Florida
  - Olympian Clinical Research, Tampa, Florida
  - The University of South Florida Board of Trustees, A public Body Corporate, for University of South Florida, Tampa, Florida
  - Northwest Behavioral Research Center, Marietta, Georgia
  - AMR - Baber Research, Inc., Naperville, Illinois
  - Psychiatric Associates, Overland Park, Kansas
  - Louisiana Clinical Research, Shreveport, Louisiana
  - Sheppard Pratt Health System, Baltimore, Maryland
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - Alivation Research, Lincoln, Nebraska
  - Healthy Perspectives - Innovative Mental Health Services. PLLC, Nashua, New Hampshire
  - Hassman Research Institute, LLC, Berlin, New Jersey
  - Global Medical Institute, LLC, Princeton, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Albuquerque Neuroscience, Inc, Albuquerque, New Mexico
  - SPRI Clinical Trials, Inc, Brooklyn, New York
  - Manhattan Behavioral Medicine, New York, New York
  - Fieve Clinical Research, New York, New York
  - New Hope Clinical Research Inc., Charlotte, North Carolina
  - Dr. Cherian Verghese, Norristown, Pennsylvania
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - Houston Clinical Trials, LLC, Bellaire, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Psychiatric and Behavioral Solutions, Salt Lake City, Utah
  - Department of Psychiatry and Neurobehavioral Sciences, University of Virginia, Charlottesville, Virginia
  - Psychiatric Alliance of the Blue Ridge, Inc., Charlottesville, Virginia

REFERENCES:
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to randomization, patients entered a 1-wk, double-blind, placebo lead-in period to identify placebo responders. Upon completion of the placebo lead-in period, patients were randomized in 1:1 ratio to receive either rapastinel or placebo. Randomization was stratified by patient's responder status (placebo non-responder vs. placebo responder).
Period: Overall Study
Arm/Group | Placebo | Rapastinel 450 mg
Started | 209 | 206
Completed | 204 | 201
Not Completed | 5 | 5
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 3 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Population: The modified Intent-to-Treat (mITT) Population will consist of all patients who were randomized, received at least 1 dose of IP during the randomized treatment period, and had at least 1 post-randomization assessment of the MADRS total score.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rapastinel 450 mg | Total
Number analyzed (Participants) | 209 | 206 | 415
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.4 (11.93) | 47.4 (11.34) | 46.9 (11.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 156 | 307
  Male | 58 | 50 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 34 | 59
  Not Hispanic or Latino | 184 | 172 | 356
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 156 | 157 | 313
  Black or African American | 48 | 45 | 93
  Asian | 3 | 3 | 6
  American Indian or Alaska Native | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
MADRS total score at baseline [Mean (Standard Deviation); unit: Scores on a Scale] — The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. Participants are rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score ranges from 0 to 60 with a higher score indicating more depression. A negative change score indicates improvement.
  Scores on a Scale | 33.8 (4.83) | 34.1 (4.73) | 34.0 (4.76)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at the End of Study
Description: The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. Participants are rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score ranges from 0 to 60 with a higher score indicating more depression. A negative change score indicates improvement.
Time Frame: Baseline and 3 Weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Rapastinel 450 mg
Number analyzed (Participants) | 209 | 206
Score on a Scale | -4.1 (0.64) | -5.1 (0.66)
Statistical Analysis 1: Comparison: Placebo vs Rapastinel 450 mg; Test type: Superiority; p = 0.2398, Mixed Model Repeated Measures (MMRM); Least Squares Mean Difference = -1.0, 95% CI 2-sided [-2.70 to 0.68]

2. Secondary Outcome: Change From Baseline in MADRS Total Score
Description: as for outcome 1
Time Frame: Baseline and Day 8
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Rapastinel 450 mg
Number analyzed (Participants) | 209 | 206
Score on a Scale | -4.3 (0.53) | -3.9 (0.55)
Statistical Analysis 1: Comparison: Placebo vs Rapastinel 450 mg; Test type: Superiority; p = 0.5522, Mixed Model Repeated Measures (MMRM); Least Squares Mean Difference = 0.4, 95% CI 2-sided [-0.95 to 1.77]

3. Secondary Outcome: Change From Baseline to Day 21 in MADRS Total Score for the Placebo Non-responders of mITT Population
Description: as for outcome 1
Time Frame: Baseline and Day 21
Population: The baseline population for placebo non-responders is 284.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Rapastinel 450 mg
Number analyzed (Participants) | 145 | 139
Score on a Scale | -4.6 (0.72) | -4.6 (0.74)
Statistical Analysis 1: Comparison: Placebo vs Rapastinel 450 mg; Test type: Superiority; p = 0.9901, Mixed Model Repeated Measures (MMRM); Least Squares Mean Difference = -0.0, 95% CI 2-sided [-2.01 to 1.99]

4. Secondary Outcome: Change From Baseline to Day 8 in MADRS Total Score for the Placebo Non-responders of mITT Population
Description: as for outcome 1
Time Frame: Baseline and Day 8
Population: The baseline population for placebo non-responders is 284.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Rapastinel 450 mg
Number analyzed (Participants) | 145 | 139
Score on a Scale | -4.1 (0.61) | -3.6 (0.62)
Statistical Analysis 1: Comparison: Placebo vs Rapastinel 450 mg; Test type: Superiority; p = 0.5563, Mixed Model Repeated Measures (MMRM); Least Squares Mean Difference = 0.5, 95% CI 2-sided [-1.17 to 2.17]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for up to 28 days.
Description: The Safety Population will consist of all patients who were randomized and received at least 1 dose of IP during the randomized treatment period.
Arm/Group | Placebo | Rapastinel 450 mg
All-Cause Mortality (participants affected / at risk) | 1/209 | 0/206
Serious Adverse Events (participants affected / at risk) | 3/209 | 0/206
Other Adverse Events (participants affected / at risk) | 18/209 | 15/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=209) | Rapastinel 450 mg (N=206)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1/151 | 0/156
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=209) | Rapastinel 450 mg (N=206)
Headache (Nervous system disorders) | 18 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT02943577/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/77/NCT02943577/SAP_001.pdf